CLINICAL TRIAL: NCT04031183
Title: Population Pharmacokinetics of Metronidazole in Neonates: Evaluation and Optimization of the Dose
Brief Title: Population Pharmacokinetics of Metronidazole in Neonates
Acronym: METROPOP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC18_8856_METROPOP
Record Dates: First submitted 2019-07-01; First posted 2019-07-24 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-03

CONDITIONS: Emergencies
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood or peritoneal fluid drawn for routine biochemical tests
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of NEOPOPI is to conduct a population pharmacokinetic study of metronidazole in neonates, in order to evaluate and optimize neonatal dose regimen.

There will be no change to the medication treatment received by participants. An opportunistic pharmacokinetic sampling approach will be followed: samples will be scavenged from blood or cerebrospinal fluid drawn for routine biochemical tests. In this way, no additional invasive tests will be needed.

DETAILED DESCRIPTION:
* Administration of the antibiotic according to the usual procedures for prescribing services: in particular, neither the indications nor the doses nor the methods of administration are fixed by the protocol
* Opportunistic sampling strategy: no biological samples are specifically collected for the purposes of the study (measurements of concentrations on "bottoms" or "left-over" samples); the performance of this non-invasive sampling strategy has been previously demonstrated in the neonatal population.
* Micro-analytical method (assay of concentrations on micro-volumes, of the order of 50μL)
* Population pharmacokinetic analysis

ELIGIBILITY:
Inclusion Criteria:

* In case of birth at gestational age ≥ 37 weeks of amenorrhea (SA): inclusion of children of postnatal age <28 days
* In case of birth at a gestational age <37 SA: inclusion of post-menstrual age children (ie gestational age + post-natal age) <44 SA 2. Benefiting from metronidazole antibiotic therapy, as part of their routine independent clinical management of the study, whether the targeted infection is suspected or proven 3. Social Security Affiliates 4. No opposition of parents to participation in the study

Non-Inclusion Critéria Treatment with metronidazole initiated before arrival in the investigative center (> 1 dose).

Exclusion Criteria:

* None

Max Age: 44 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates (including both preterm and full-term neonates) receiving amoxicillin as part of their routine clinical care (for suspected or proven neonatal sepsis).
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2020-05-29 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Achievement rate of therapeutic efficacy target of metronidazole | 1 week
  Achievement rate of therapeutic efficacy target of Metronidazole (ie percentage of neonates in whom metronidazole plasma concentration remains above the MIC of target organisms for more than 70% of the dose range). In accordance with the recommendations of the European Medicines Agency, the optimal dosage regimen is defined as leading to a probability of antibiotic therapy success of greater than or equal to 90%. Thus, it is necessary to determine the dosage regimen allowing the target of therapeutic efficacy to be reached (ie maintenance of the plasma concentration of metronidazole greater than the MIC of the targeted microorganisms for more than 70% of the dose) in at least 90% of treated neonates.

SECONDARY OUTCOMES:
Number of Adverse Events | 1 week
  Recording of adverse events (clinical and / or biological) during the treatment period and up to the end of the hospitalisation
Minimum Inhibitory Concentration | 1 week
  Collection of MICs of metronidazole for isolated germs. For metronidazole the antibacterial activity is time-dependent, the predictor of efficacy is the "Time> MIC": this is the percentage of the administration interval during which the concentration of the antibiotic remains higher than the MIC of target germs
Concentration of metronidazole un peritoneal fluid | 1 week
  Calculation of metronidazole concentration in peritoneal fluid / metronidazole plasma concentration when data permits (i.e. when prelevment performed as part of usual care, during treatment with metronidazole
average clearance | 1 week
  Using the population pharmacokinetic model developed and validated (diagnostic plots, NPDE (Comets et al., 2008), and bootstrap), calculation of:
  - the precision of estimates of average clearance
Impact of age | 1 week
  Using the population pharmacokinetic model developed and validated (diagnostic plots, NPDE (Comets et al., 2008), and bootstrap), calculation of:
  the impact of âge associations as explaining part of the pharmacokinetic variability of the antibiotic
Impact of weight | 1 week
  Using the population pharmacokinetic model developed and validated (diagnostic plots, NPDE (Comets et al., 2008), and bootstrap), calculation of:
  the impact of weight as explaining part of the pharmacokinetic variability of the antibiotic
Impact of therapeutic associations | 1 week
  Using the population pharmacokinetic model developed and validated (diagnostic plots, NPDE (Comets et al., 2008), and bootstrap), calculation of:
  the impact of therapeutic associations as explaining part of the pharmacokinetic variability of the antibiotic
volume of distribution | 1 week
  Using the population pharmacokinetic model developed and validated (diagnostic plots, NPDE (Comets et al., 2008), and bootstrap), calculation of:
  - the precision of estimates of volume of distribution
interindividual variability | 1 week
  Using the population pharmacokinetic model developed and validated (diagnostic plots, NPDE (Comets et al., 2008), and bootstrap), calculation of:
  - the precision of estimates of interindividual variability
residual variability | 1 week
  Using the population pharmacokinetic model developed and validated (diagnostic plots, NPDE (Comets et al., 2008), and bootstrap), calculation of:
  - the precision of estimates of residual variability

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - CHU d'Angers, Angers
  - CHU de Brest, Brest
  - Centre Robert Debré, Paris
  - CHU de Rennes, Rennes
  - CH St Brieuc, Saint-Brieuc
  - CHU de Tours, Tours
  - CH Vannes, Vannes